CLINICAL TRIAL: NCT03150355
Title: Outcomes of Geriatric Hip Fractures in Assiut University Hospital
Status: Completed | Type: Observational
Sponsor: khaled (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, khaled, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: khaled38
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Arthroplasty; Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- open reduction and internal fixation: outcome of open reduction and internal fixation of fractures of proximal femur and acetabulum in patients aged 65 years and older
  Interventions: Procedure: Arthroplasty or open reduction and internal fixation
- Arthroplasty: outcome of arthroplasty of fractures of proximal femur and acetabulum in patients aged 65 years and older
  Interventions: Procedure: Arthroplasty or open reduction and internal fixation
- conservative management: outcome of conservative management of fractures of proximal femur and acetabulum in patients aged 65 years and older

INTERVENTIONS:
Procedure: Arthroplasty or open reduction and internal fixation — fixation of proximal femoral fractures or replacement with prosthesis
  Groups: Arthroplasty; open reduction and internal fixation

SUMMARY:
hip fractures are common problem specially in elderly population the incidence is increasing nowadays because of increased incidence of motor vehicle accidents

DETAILED DESCRIPTION:
hip fractures are a common problem specially in elderly population the incidence is increasing nowadays because of increased incidence of motor vehicle accidents the incidence of morbidity and mortality is increasing today and the mortality rate is about 30% the aim of the study is follow up of the patients aged 65 years and older who experienced hip fractures for one year to evaluate the outcome of different ways of intervention in elderly population.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years and older
* with fractures acetabulum , neck of femur , trochanteric , subtrochanteric and reverse trochanteric fractures

Exclusion Criteria:

* no patient will be excluded

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged 65 years old and older with fracture acetabulum , neck of femur , trochanteric , subtrochanteric and reverse trochanteric fractures admitted inside assuit university hospital
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
determine the outcome of geriatric hip fractures | one year
  determine the morbidity and mortality of surgery of hip fractures in elderly patients aged 65 years and older

SECONDARY OUTCOMES:
determine magnitude of geriatric hip fractures | one year
  determine incidence of hip fractures which is increasing nowadays

OTHER OUTCOMES:
determine the readmission rate to the hospital and why they were readmitted | one year
  determine the readmission rate to the hospital and why they were readmitted to the hospital due to metal failure , infection ...etc
determine the risk factors for morbidity and mortality | one year
  determine what are the factors and causes that increase the risk of morbidity and mortality in the patients

IPD SHARING:
Plan to Share IPD: No